CLINICAL TRIAL: NCT06046066
Title: A Phase I Study to Determine the Maximum Tolerated Dose and Evaluate Safety, Tolerability, and Pharmacokinetics of NM6603 in Patients With Advanced Solid Tumors
Brief Title: A Phase 1 Study of NM6603 in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NucMito Pharmaceuticals Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NM6603-CP-101
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-03

CONDITIONS: Cancers
Keywords: advanced solid tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): NM6603, administered orally every day in 28-day cycles
  Interventions: Drug: NM6603

INTERVENTIONS:
Drug: NM6603 — NM6603 is an orally available investigational small molecule indicated for the treatment of solid malignancies including, but not limited to breast, liver, pancreatic, colorectal, cervical, melanoma and lung cancers.

SUMMARY:
This study is to assess the MTD and RP2D of NM6603 in adult patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1, first-in-human, multicenter, open label, 3+3 dose escalation study designed to evaluate the safety profile, the maximum tolerated dose (MTD), the recommended Phase 2 dose (RP2D), the pharmacokinetic and the preliminary antitumor activity of NM6603 in patients with advanced solid tumors. The study has two parts. In Part 1, NM6603 will be administered once daily. In Part 2, NM6603 will be administered twice daily to explore the effect of twice daily dosing on the pharmacokinetic, safety and tolerability, and anti-tumor activity profile of NM6603,

ELIGIBILITY:
Inclusion Criteria:

1. Have a histologically or cytologically confirmed diagnosis of advanced solid tumor;
2. Have advanced or metastatic disease refractory to standard curative or palliative therapy or contraindication to standard therapy;
3. Have objective (assessable through clinical signs, symptoms, and/or laboratory findings) and radiologically-confirmed progression of disease at Screening;
4. Patients must have measurable disease based on RECIST v1.1;
5. ≥ 18 years of age;
6. Patients must exhibit a/an ECOG performance status of 0-2;
7. Have a life expectancy of at least 12 weeks (in the opinion of the investigator);
8. Have adequate bone marrow reserve:

   1. Absolute neutrophil count ≥1.5×109 cell/L;
   2. Platelet count ≥100×109 cell/L;
   3. Hemoglobin at least ≥9.0 g/dL
9. Have adequate liver function:

   1. Total serum bilirubin ≤ 1.5× upper limit of normal (ULN);
   2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5× ULN or ≤5.0× ULN in case of documented hepatic metastasis;
   3. Alkaline phosphatase ≤ 5× ULN
10. Have adequate renal function:

    1. glomerular filtration rate ≥60 mL/min (calculated according to the formula of Cockcroft and Gault);
    2. No clinically relevant abnormalities in the urinalysis results
11. Are capable of swallowing study medication and following directions regarding taking study drug;
12. Women of childbearing potential (WOCBP) and Women of non-childbearing potential are eligible to participate. Both women of childbearing potential and women of non-childbearing potential should use an approved method of birth control and agrees to continue to use this method for the duration of the study and for 90 days after taking the last dose of study drug.

    Acceptable methods of contraception include abstinence, female subject/partner's use of hormonal contraceptive (oral, implanted, or injected) in conjunction with a barrier method (WOCBP only) (e.g., diaphragm, cervical cap, male condom, and female condom and spermicidal foam, sponges, and film), female subject/partner's use of an intrauterine device (IUD), or if the female subject/partner is surgically sterile (e.g., bilateral tubal ligation, hysterectomy) for at least 3 months before screening or two years postmenopausal at time of screening. All male subjects/partners (excluding men who have been sterilized) must agree to consistently and correctly use a condom for the duration of the study and for 90 days after taking the study drug. In addition, subjects may not donate sperm for the duration of the study and for 90 days after taking study drug.

    Note: Women of non-childbearing potential who are less than two years postmenopausal should be tested for pregnancy. Any verbal confirmation of postmenopausal status will be recorded in source documents and appropriate page of CRF.
13. WOCBP must have a negative serum pregnancy test at Screening Visit and negative urine pregnancy test prior to receiving the first dose of study drug; and
14. Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study.

Exclusion Criteria: Subjects meeting any of the following criteria will be excluded from enrollment:

1. Have unresolved toxicity from previous treatment or previous investigational agents, excluding alopecia. Clinical judgment by the investigator is allowed to determine if grade 1 fatigue at screening is residual toxicity from prior treatment or is a symptom of the patient's general condition or disease or if > Grade 1 toxicities are non-clinically relevant such as Lymphopenia. The investigator and medical monitor will discuss the eligibility of patients with baseline toxicity;
2. Have signs or symptoms of end organ failure, major chronic illnesses other than cancer, or any severe concomitant conditions which, in the opinion of the investigator, make it undesirable for the patient to participate in the study, or which could jeopardize compliance with the protocol;
3. Have evidence of another malignancy not in remission or history of such a malignancy within the last three years (except for treated basal or squamous cell carcinoma of the skin, or in situ cancer of the cervix);
4. Have abnormalities in the 12-lead ECG that in the opinion of the Investigator increase the risk of participating in the study (e.g., sinus rhythm with PR interval > 240 ms or second degree or higher AV block, confirmed by a repeat ECG);
5. Have ECG evidence of complete left bundle branch block or ventricular pacing;
6. Have a history of long QT syndrome or prolonged QT interval corrected based on Fridericia's method (QTcF) >450 ms at screening;
7. Require treatment with drugs known to be associated with Torsade de Pointes;
8. Have experienced any of the following within the 6-month period prior to screening that would interfere with the subject's participation in the opinion of the treating investigator: unstable angina, myocardial infarction or cerebrovascular accident, transient ischemic attack, cardiac failure with known ejection fraction less than 40%;
9. Have other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that would make the patient inappropriate for enrollment in this study;
10. Have any mental or medical condition that prevents the subject from giving informed consent or participating in the trial;
11. Have received anti-tumor therapies such as chemotherapy, hormone therapy, radiation therapy, or immunotherapy within 4 weeks or 4 half-lives (whichever is shorter or as agreed between the site PI and Medical Monitor) prior to starting the study drug;
12. Have received systemic corticosteroids (either oral or intravenous steroids, excluding inhalers or topicals) for a duration ≥ 4 weeks at the daily dose equivalent to ≥7.5 mg of oral prednisone within the 12 weeks prior to starting study drug;
13. Are currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 28 days or four half-lives (whichever is shorter, or as agreed between the site PI and Medical Monitor) prior to first study drug administration;
14. Have known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Note: Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability;
15. Require treatment with strong inhibitors, strong inducers, and/or sensitive substrates of CYP1A2 and/or CYP3A4, and/or sensitive substrates of CYP2B6 or major drug transporters; This medication can be stopped and the patient enrolled after 4 half- lives of that drug, as determined by the PI.
16. Are unwilling to or unable to comply with the requirement of the protocol; and
17. Are pregnant or breastfeeding or expecting to conceive or have children within the projected duration of the trial, starting with the pre-screening or screening visit through the duration of study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and recommended Phase II dose (RP2D) of NM6603 in patients with advanced solid tumors | 28 days

SECONDARY OUTCOMES:
Efficacy of NM6603 by Objective Response Rate (ORR) via iRECIST | From first dose of study drug to up to ~ 12 months in absence of progressive disease or unacceptable toxicity or withdrawal of consent
Efficacy of NM6603 by disease control rate (DCR) via iRECIST | From first dose of study drug to up to ~ 12 months in absence of progressive disease or unacceptable toxicity or withdrawal of consent
Pharmacokinetics (PK) of NM6603 by maximum observed plasma drug concentration (Cmax) | 28 days
Pharmacokinetics (PK) of NM6603 by apparent terminal elimination half-life (t1/2) | 28 days
Pharmacokinetics (PK) of NM6603 by time to maximum observed plasma drug concentration (Tmax) | 28 days
Pharmacokinetics (PK) of NM6603 by area under the plasma drug concentration-time curve (AUC) from time 0 to the time of the last quantifiable concentration (Tlast) (AUC0-t) | 28 days
Pharmacokinetics (PK) of NM6603 by AUC from time 0 to infinity (AUC0-∞) | 28 days
Safety of NM6603 by Dose-Limiting Toxicities | 28 days
Safety of NM6603 by incidence and severity of treatment-emergent adverse events (TEAEs) | From first dose of study drug to up to ~ 12 months in absence of progressive disease or unacceptable toxicity or withdrawal of consent
  The intensity of the event will be graded using CTCAE v5.0 criteria.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Karmanos Cancer Institute, Detroit, Michigan
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No